CLINICAL TRIAL: NCT06698133
Title: Knowledge and Habits of Pregnant Teens: Analyzing Nutritional Status, Weight and Infant Birth Weight
Brief Title: Knowledge and Habits of Pregnant Teens
Acronym: KnowTeens
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Sheila Belk, Assistant Professor, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UMMC IRB 2024-447; pending (Other: pending)
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Teen Pregnancy
Keywords: Gestational Weight Gain; Infant Birth Weight; Health Literacy
MeSH Terms: conditions — Gestational Weight Gain

STUDY DESIGN:
Intervention Model Description: Participants in the intervention arm will be invited to join a private social media group that will be created solely for this study. Education content will consist of published dietary recommendations during pregnancy, healthy craving hacks, healthy snacks, ways to get exercise in during the school day, etc. Participants will also be encouraged to ask questions and post any eating struggles. The intervention will be completely virtual and outside of the initial visit. Medical advice will not be given; if requested, participants will be advised to contact their provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (No Intervention): Control Group will complete the 20 questions health literacy during the first visit and after 8 weeks. Also, will complete the online called ASA 24 a 24-hour food recall tool. The ASA24 will be completed 2x /week for 8 weeks.
- Intervention Arm (Experimental): Intervention Group will complete the 20 questions health literacy during the first visit and after 8 weeks. Also, will complete the online called ASA 24 a 24-hour food recall tool. The ASA24 will be completed 2x /week for 8 weeks. In addition, participants assigned to the intervention group will be invited to participate in a private social media group.
  Participants in the intervention arm will be invited to join a private social media group that will be created solely for this study. This will be a private account, accessible only to participants who are added or invited by the study team.
  Interventions: Other: Participants in the intervention arm will be invited to join a private social media group

INTERVENTIONS:
Other: Participants in the intervention arm will be invited to join a private social media group — Education content
  Arms: Intervention Arm

SUMMARY:
This study examines the link between health literacy, gestational weight gain, and infant birthweight in pregnant teenagers. A randomized trial of 50 participants will be conducted at the University of Mississippi Medical Center. Consent will be obtained from all participants. Both control and intervention groups will complete a 20 questions health literacy assessment at baseline and after eight weeks, along with the ASA24 dietary recall tool twice weekly. The intervention group will join a private social media group created solely for study purposes. This will be a private account, accessible only to participants who are added or invited by the study team.

DETAILED DESCRIPTION:
This research study is to see if someone's ability to understand and use health information (health literacy) is linked to gaining a healthy amount of weight during pregnancy and having a baby with a healthy birth weight. The main question aims to answer if there is a positive correlation between increased health literacy, gestational weight gain, and adequate infant birth weight. We are conducting a prospective randomized trial involving 50 pregnant teenagers and their baby at a single institution. We will obtain study consent for 18 and 19 years old, and parental permission and assent for 13 -17 years old.

Control Group will complete the 20 questions health literacy during the first visit and after 8 weeks. Also, will complete the online called ASA 24 a 24-hour food recall tool. The ASA24 will be completed 2x /week for 8 weeks.

Intervention Group will complete the 20 questions health literacy during the first visit and after 8 weeks. Also, will complete the online called ASA 24 a 24-hour food recall tool. The ASA24 will be completed 2x /week for 8 weeks. In addition, participants assigned to the intervention group will be invited to participate in a private social media group. Participants will create a new account specifically for the study, or the study team can create an account on their behalf if they prefer. This will enable the study team to track participation without affecting any personal accounts. Education content will consist of published dietary recommendations during pregnancy, healthy craving hacks, healthy snacks, ways to get exercise in during the school day, etc. Participants will also be encouraged to ask questions and post any eating struggles.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age 13 - 19 yrs at enrollment
* < 19.6 gestational weeks
* Ability to understand English
* Access to a smartphone or internet
* Willingness to follow study procedures
* Plan to deliver at UMMC
* Singleton pregnancy

Exclusion Criteria:

* Does not meet the inclusion criteria
* History of diabetes
* Current record of substance abuse
* Mental impairment
* Eating disorder

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Health Literacy | All study participants will complete this survey at the beginning of the study and again after week 8.
  All data collected in the study design will be used to answer questions in this aim. The Maternal Health Literacy (MaHeLi) is a 20-item questionnaire used to assess health literacy in adolescents .

SECONDARY OUTCOMES:
Demographic Information | From enrollment to the end of 8 weeks
  Demographic information will be collected, such as maternal age, gender, race, pre-pregnancy body mass index, weight, height, and BMI. Obstetrical and medical history will also be collected but not limited to gestational age, historical and current maternal outcome. Infant data will also be collected, such as gender, birth weight, infant unit admission, and infant outcome.

OTHER OUTCOMES:
24-hour food recall tool | The ASA24 will be completed 2x /week for 8 weeks.
  All study participants must complete the Automated Self-Administered 24-hour (ASA24) Dietary Assessment Tool to record dietary intakes. The ASA24 dietary assessment tool is a web-based tool designed for collecting detailed dietary intake information. ASA24 allows researchers and individuals to obtain dietary data through a 24-hour recall process, where participants report all the foods and beverages they consumed in the past 24 hours. ASA24 uses a large database of foods, providing nutritional information like calories, macronutrients, vitamins and minerals.

IPD SHARING:
Plan to Share IPD: No